CLINICAL TRIAL: NCT02394977
Title: Pilot Study of the Effect of Cardio First Angel (CFA) Device on CPR Outcomes:
Brief Title: Effect of the Cardio First Angle Device on CPR Outcomes
Acronym: CFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other); West Virginia University (Other)
Responsible Party: Principal Investigator, Amir Vahedian-Azimi, Senior intensivist nurse, Respiratory therapist, Research Fellow, PhD, RN, FCCS, Baqiyatallah Medical Sciences University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: BMSU-390-5-5904
Record Dates: First submitted 2015-03-05; First posted 2015-03-20 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Cardiopulmonary Arrest
Keywords: CPR; Cardio first angle; Clinical trial
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Compression with Feedback (Experimental): CPR performed according to established international standards with chest compressions performed with the assistance of the Cardio First Angel™ (CFA; INOTECH, Nubberg, Germany) compression feedback device.
  Interventions: Device: Compression with Feedback
- Standard chest compression (Active Comparator): CPR performed according to established international standards with standard manual chest compression
  Interventions: Other: Standard chest compression

INTERVENTIONS:
Device: Compression with Feedback — Patients in the intervention group received CPR in accordance to published guidelines using the CFA device per manufacturer instructions. The Cardio First Angel™ (CFA; INOTECH, Nubberg, Germany) is a lightweight device that consists of three components . Application of400 ± 30 Newtons of force (41 kg or 90 lb of pressure), which correlates toa sternum compression depth of 50-60 mm, is followed by an audible "click" sound to alert the rescuer to cease compression. The "click" sound is also audible upon spring decompression alerting the rescuer to resume compression. The device does not require an electrical power supply.
  Other Names: Cardio First Angel™
  Arms: Compression with Feedback
Other: Standard chest compression — CPR in accordance with published international guidelines using standard manual chest compression.
  Arms: Standard chest compression

SUMMARY:
The investigators conducted a randomized, controlled, single-blinded study of patients undergoing CPR for cardiac arrest in the mixed medical-surgical ICUs of four academic teaching hospitals in Tehran, Iran from June 1 to October 31, 2014. Patients were randomized to receive CPR with either standard manual compression, or compression with real-time audiovisual feedback using the Cardio First Angel™ device.

DETAILED DESCRIPTION:
The investigators sought to determine if the addition of a CPR feedback device to routine manual CPR would impact the quality and consistency of chest compression and patient survival. We conducted a randomized, controlled, single-blinded study of patients undergoing CPR for cardiac arrest in the mixed medical-surgical ICUs of four academic teaching hospitals. Patients were randomized to receive either standard manual CPR or CPR using the Cardio First Angel™ (CFA; INOTECH, Nubberg, Germany) feedback device. Recorded variables included return of spontaneous circulation, adherence to CPR guidelines and quality of CPR, nurse satisfaction and CPR associated morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admitted to the intensive care unit (ICU)
* Full-code status
* Informed consent was obtained from the patient, legal guardian, or healthcare surrogate upon ICU admission (prior to cardiac arrest event)

Exclusion Criteria:

* Patients with any limitation of code status including but not limited to "no code" or"do not resuscitate" (DNR) and"do not intubate" (DNI), were excluded from study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Sustained Return of Spontaneous Circulation | through resuscitation completion, an average of 30 to 60 minutes
  ROSC lasting > 30 minutes

SECONDARY OUTCOMES:
Nurse Satisfaction Score | upon resuscitation completion, an average of 30 to 60 minutes
  Nurse satisfaction with resuscitation event using a validated tool
CPR Duration | through resuscitation completion, an average of 30 to 60 minutes
  Duration of CPR event
New post-resuscitation Sternum or Rib Fractures | through resuscitation completion, an average of 30 to 60 minutes
  New sternum or Rib Fractures diagnosed post-resuscitation using X-ray, CT scan, or by Autopsy
CPR Evaluation Score | upon resuscitation completion, an average of 30 to 60 minutes
  CPR evaluation score assess quality of CPR including chest compression sing a validated tool
CPR Guideline Observation Score | upon resuscitation completion, an average of 30 to 60 minutes
  Assesses guideline adherence

CONTACTS AND LOCATIONS:
Overall Officials: Amir vahedian-azimi, PhD, RN, Principal Investigator — BMSU

REFERENCES:
- [Result] Vahedian-Azimi A, Hajiesmaeili M, Amirsavadkouhi A, Jamaati H, Izadi M, Madani SJ, Hashemian SM, Miller AC. Effect of the Cardio First Angel device on CPR indices: a randomized controlled clinical trial. Crit Care. 2016 May 17;20(1):147. doi: 10.1186/s13054-016-1296-3. PMID 27184664
- See also: "Critical Care" site for full text — http://ccforum.biomedcentral.com/articles/10.1186/s13054-016-1296-3#Sec11